CLINICAL TRIAL: NCT03097146
Title: Managing Aftercare for Stroke (MAS): MAS-II - A Longitudinal Complex-interventional Study in Post-rehabilitation Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Stroke Research Berlin (Other); Hebrew University of Jerusalem (Other); NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MAS-II
Record Dates: First submitted 2017-03-27; First posted 2017-03-31 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Stroke
Keywords: Stroke; Aftercare; Comprehensive Care
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- comprehensive multidisciplinary stroke care (Other)
  Interventions: Other: comprehensive multidisciplinary stroke care

INTERVENTIONS:
Other: comprehensive multidisciplinary stroke care — Patients will be treated in the pathological domain. Some of this treatment will be applied by the outpatient clinic itself (i.e. changes in medical secondary prevention or additional prescriptions, social work interventions), whereas most of it will be referred to other providers, if possible in vicinity to the patients' home. In order to ease treatment prescriptions and allow to measure treatment uptake, patients will also enrol in the case management system "Ambulanzpartner". This allows the outpatient center to streamline prescription processes and measure uptake of therapies.

SUMMARY:
After discharge from hospital, the current healthcare system in Germany allows considerable flexibility (therefore complexity) of patient access and mobility between multiple care providers in the community setting. The investigators believe this aftercare could be better coordinated by a specialized coordinated stroke aftercare service. Comprehensive coordinated multidisciplinary care is a proven concept with proven benefits in both acute and rehabilitation care provided in stroke units and neurorehabilitation centres. In this study, the investigators postulate that a similar coordinated approach to care can be extended to the phase after in-patient rehabilitation has ended (i.e. "long-term management" as opposed to "early supported discharge") for disabled patients with stroke living in the community.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke
* Age ≥18 years
* At the time of V1 completion of rehabilitation or no rehabilitation planned
* Informed consent signed by patient or legal representative
* stroke patients with a stratified mRS score
* within six months after the index event

Exclusion Criteria:

* Unwillingness to participate in "AmbulanzPartner"
* Unwilling to have pseudonymized data stored, analysed, and anonymously published
* Patients being committed to psychiatric institutions or prisons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
"EuroQol five dimensions questionnaire" (EuroQoL-5D) | 12 Months
  questionnaire for self-completion by patients for use as a measure of health outcome

SECONDARY OUTCOMES:
Post Stroke Checklist (PSC) | 12 Months
  checklist that helps identify post-stroke problems
modified Rankin Scale (mRS) | 12 Months
  scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability
Barthel-Index (BI) | 12 Months
  scale is used to measure performance in activities of daily living
modified Ashworth Scale (mAS) | 12 Months
  scale is used as a measure of spasticity
Pain Detect (PD-Q) | 12 Months
  questionnaire for self-completion by patients for the identification of neuropathic pain
Freiburg questionnaire for coping (FKV) | 12 Months
  questionnaire is used to assess disease processing modes at the levels of cognition, emotion, and behavior
Montreal Cognitive Assessment (MoCA) | 12 Months
  cognitive screening test in the detection of mild cognitive impairment
partial Aachen Aphasia Test (AAT) | 12 Months
  test is used to diagnose and describe aphasic disturbances
Hamilton rating scale for depression | 12 Months
  questionnaire is used to provide an indication of depression
"Morisky Medication Adherence Scale" (MMAS) | 12 Months
  questionnaire is used to assess patients' medication-taking behaviour
"Nikolaus score for evaluation of social conditions" (SoS) | 12 Months
  score is used to assess patients' social work intervention
"Häusliche Pflegeskala" (HPS) | 12 Months
  questionnaire is used to assess social work Intervention and couple's counselling
Hospital Anxiety Depression Scale (HADS) | 12 Months
  questionnaire for self-completion by patients to determine the levels of anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- NeuroCure Clinical Research Center (NCRC), Charité, Berlin, Germany